CLINICAL TRIAL: NCT03441685
Title: Strategies for Teaching Verbs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Melanie Schuele, Associate Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 172058
Record Dates: First submitted 2018-02-08; First posted 2018-02-22 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2023-12

CONDITIONS: Language Development Disorders; Down Syndrome; Child Language
MeSH Terms: conditions — Language Development Disorders; Down Syndrome

STUDY DESIGN:
Intervention Model Description: All participants complete the three intervention conditions within a single session. Order of conditions is counterbalanced across participants.
Masking Description: Participants' completion of study tasks requires knowledge of intervention condition. Participants are blinded to study hypotheses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Verb strategies (Experimental): The examiner labels each target word and performs the corresponding action six times in each condition. She elicits the target word from the participant two times per word per condition and provides feedback on accuracy each time. In the semantic cues condition, the examiner prompts the child to perform the target action twice. In the syntactic cues condition, instead of only saying the target word with the present progressive verb marker, the examiner uses two forms of complete sentences while performing the action (i.e., "I am X-ing," and "See. I X."). In the combined condition, the examiner prompts the child to perform the target action and consistently uses complete sentences.
  Interventions: Behavioral: Semantic cues (perform action), syntactic cues (sentence frame), or combined semantic and syntactic cues

INTERVENTIONS:
Behavioral: Semantic cues (perform action), syntactic cues (sentence frame), or combined semantic and syntactic cues — Verb Learning Session Teaching phase. The examiner labels each target word and performs the action 6 times in each condition. She elicits the target word from the participant 2 times per word per condition and provides feedback on accuracy.
  Testing phase. Receptive probes are administered after every 2 words are taught. Expressive probes are at the end of the condition. For receptive probes, the examiner asks the participant to identify novel verbs and for expressive probes, the examiner asks the child to label the novel action. Testing after 2 items is designed to decrease memory load. Participants have a brief break between conditions.
  Data are collected on: a) child responses on standardized assessments, (b) responses to verb learning probes, (c) parent responses to intake form, and (d) relevant medical history from electronic medical record.
  None of the above procedures present more than minimal risk to participants or research staff. Vanderbilt IRB approved all procedures.

SUMMARY:
This study is designed to evaluate whether children with Down syndrome and children with typical development exhibit different levels of accuracy demonstrating novel verbs taught under three conditions: semantic cues (perform action), syntactic cues (sentence frame), and combined (syntactic and semantic cues). The participants complete an eligibility evaluation and then one verb learning session (approximately 60 minutes in length). During that verb learning session they are taught sets of words under each condition (i.e., within-subjects design) and then asked to identify and label those target words immediately after instruction.

ELIGIBILITY:
Inclusion Criteria:

* Must use oral communication as their primary means of communication
* Must be monolingual English speakers
* Behaviorally able to attend for 20 minutes
* Children with typical development must demonstrate no more than one standard deviation below the mean on the speech and language measures

Exclusion Criteria:

* Nonverbal cognitive score less than three standard deviations below the mean (standard score of 54 below)
* Identified hearing loss or failed hearing screening
* Uncorrected vision impairment
* Motor impairment that prevents completion of study activities
* Concomitant disorders (e.g., Autism spectrum disorder)

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt Bill Wilkerson Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Typical Development: Children with typical development
- Down Syndrome: Children with Down syndrome
- Developmental Language Disorder: Children with developmental language disorder
Period: Overall Study
Arm/Group | Typical Development | Down Syndrome | Developmental Language Disorder
Started | 23 | 8 | 7
Completed | 23 | 8 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Typical Development | Down Syndrome | Developmental Language Disorder | Total
Number analyzed (Participants) | 23 | 8 | 7 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 8 | 7 | 38
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 2 | 21
  Male | 10 | 2 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 3 | 5
  Not Hispanic or Latino | 20 | 7 | 4 | 31
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 17 | 8 | 4 | 29
  More than one race | 6 | 0 | 0 | 6
  Unknown or Not Reported | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 23 | 8 | 7 | 38

OUTCOME MEASURES:

1. Primary Outcome: Accuracy Identifying Taught Words - Syntactic Condition
Description: Participants are asked to receptively identify novel verbs taught in syntactic condition by selecting the video of the named verb from a field of two. Participants were asked to identify each of the 4 taught words per condition 3 times for a total of 12 trials per condition. This "receptive probe" has a minimum score of 0 and maximum of 12. Higher scores indicate a better outcome.
Time Frame: From date of initial evaluation to focused intervention session, up to 1 month
Population: Analyzed eligible participants
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Typical Development | Down Syndrome | Developmental Language Disorder
Number analyzed (Participants) | 23 | 8 | 7
Score on a scale | 8.73 (3.26) | 8.75 (3.11) | 10.29 (2.21)
Statistical Analysis 1: Comparison: Typical Development; Test type: Other — Accuracy identifying taught verbs in syntactic vs semantic condition (receptive); p = 0.73, Wilcoxon Signed Ranks Test — Asymptotic p-value
Statistical Analysis 2: Comparison: Down Syndrome; Test type: Other — Accuracy identifying taught verbs in syntactic vs semantic condition (receptive); p = 0.69, Wilcoxon Signed Ranks Test — Asymptotic p-value
Statistical Analysis 3: Comparison: Developmental Language Disorder; Test type: Other — Accuracy identifying taught verbs in syntactic vs semantic condition (receptive); p = 0.79, Wilcoxon Signed Ranks Test — Asymptotic p-value
Statistical Analysis 4: Comparison: Typical Development; Test type: Other — One-sample Wilcoxon signed rank test with comparison value of 6; p = 0.002, One-sample Wilcoxon signed rank test — Asymptotic p-value
Statistical Analysis 5: Comparison: Down Syndrome; Test type: Other — One-sample Wilcoxon signed rank test with comparison value of 6; p = 0.049, One-sample Wilcoxon signed rank test — Asymptotic p-value
Statistical Analysis 6: Comparison: Developmental Language Disorder; Test type: Other — One-sample Wilcoxon signed rank test with comparison value of 6; p = 0.016, One-sample Wilcoxon signed rank test — Asymptotic p-value

2. Primary Outcome: Accuracy Identifying Taught Words - Semantic Condition
Description: Participants are asked to receptively identify novel verbs taught in semantic condition by selecting the video of the named verb from a field of two. Participants were asked to identify each of the 4 taught words per condition 3 times for a total of 12 trials per condition. This "receptive probe" has a minimum score of 0 and maximum of 12. Higher scores indicate a better outcome.
Time Frame: From date of initial evaluation to focused intervention session, up to 1 month
Population: Analyzed eligible participants
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Typical Development | Down Syndrome | Developmental Language Disorder
Number analyzed (Participants) | 23 | 8 | 7
Score on a scale | 8.91 (3.54) | 9.50 (2.93) | 10.14 (2.67)
Statistical Analysis 1: Comparison: Typical Development; Test type: Other — Accuracy identifying taught verbs in semantic vs combined condition (receptive); p = 0.76, Wilcoxon Signed Ranks Test — Asymptotic p-value
Statistical Analysis 2: Comparison: Down Syndrome; Test type: Other — Accuracy identifying taught verbs in semantic vs combined condition (receptive); p = 0.79, Wilcoxon Signed Ranks Test — Asymptotic p-value
Statistical Analysis 3: Comparison: Developmental Language Disorder; Test type: Other — Accuracy identifying taught verbs in semantic vs combined condition (receptive); p = 1.00, Wilcoxon Signed Ranks Test — Asymptotic p-value
Statistical Analysis 4: Comparison: Typical Development; Test type: Other — One-sample Wilcoxon signed rank test with comparison value of 6; p = 0.003, One-sample Wilcoxon signed rank test — Asymptotic p-value
Statistical Analysis 5: Comparison: Down Syndrome; Test type: Other — One-sample Wilcoxon signed rank test with comparison value of 6; p = 0.029, One-sample Wilcoxon signed rank test — Asymptotic p-value
Statistical Analysis 6: Comparison: Developmental Language Disorder; Test type: Other — One-sample Wilcoxon signed rank test with comparison value of 6; p = 0.027, One-sample Wilcoxon signed rank test — Asymptotic p-value

3. Primary Outcome: Accuracy Identifying Taught Words - Combined Condition
Description: Participants are asked to receptively identify novel verbs taught in combined condition by selecting the video of the named verb from a field of two. Participants were asked to identify each of the 4 taught words per condition 3 times for a total of 12 trials per condition. This "receptive probe" has a minimum score of 0 and maximum of 12. Higher scores indicate a better outcome.
Time Frame: From date of initial evaluation to focused intervention session, up to 1 month
Population: Analyzed eligible participants
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Typical Development | Down Syndrome | Developmental Language Disorder
Number analyzed (Participants) | 23 | 8 | 7
Score on a scale | 9.04 (2.75) | 9.38 (2.07) | 10.00 (2.24)
Statistical Analysis 1: Comparison: Typical Development; Test type: Other — Accuracy identifying taught verbs in syntactic vs combined condition (receptive); p = 0.72, Wilcoxon Signed Ranks Test — Asymptotic p-value
Statistical Analysis 2: Comparison: Down Syndrome; Test type: Other — Accuracy identifying taught verbs in syntactic vs combined condition (receptive); p = 0.46, Wilcoxon Signed Ranks Test — Asymptotic p-value
Statistical Analysis 3: Comparison: Developmental Language Disorder; Test type: Other — Accuracy identifying taught verbs in syntactic vs combined condition (receptive); p = 0.89, Wilcoxon Signed Ranks Test — Asymptotic p-value
Statistical Analysis 4: Comparison: Typical Development; Test type: Other — One-sample Wilcoxon signed rank test with comparison value of 6; p < .001, One-sample Wilcoxon signed rank test — Asymptotic p-value
Statistical Analysis 5: Comparison: Down Syndrome; Test type: Other — One-sample Wilcoxon signed rank test with comparison value of 6; p = 0.018, One-sample Wilcoxon signed rank test — Asymptotic p-value
Statistical Analysis 6: Comparison: Developmental Language Disorder; Test type: Other — One-sample Wilcoxon signed rank test with comparison value of 6; p = 0.027, One-sample Wilcoxon signed rank test — Asymptotic p-value

4. Secondary Outcome: Accuracy Labeling Taught Words - Syntactic Condition
Description: After the teaching episodes for the syntactic condition participants are asked to label novel verbs expressively. Participants were asked to label each of the 4 taught words per condition one time for a total of 4 trials per condition. This "expressive probe" has a minimum score of 0 and maximum of 4. Higher scores indicate a better outcome.
Time Frame: From date of initial evaluation to focused intervention session, up to 1 month
Population: Analyzed eligible participants
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Typical Development | Down Syndrome | Developmental Language Disorder
Number analyzed (Participants) | 23 | 8 | 7
Score on a scale | 0.61 (0.58) | 0.75 (0.71) | 0.86 (0.90)
Statistical Analysis 1: Comparison: Typical Development; Test type: Other — Accuracy labeling taught verbs in syntactic vs semantic condition (expressive); p = 0.64, Wilcoxon Signed Ranks Test — Asymptotic p-value
Statistical Analysis 2: Comparison: Down Syndrome; Test type: Other — Accuracy labeling taught verbs in syntactic vs semantic condition (expressive); p = 0.16, Wilcoxon Signed Ranks Test — Asymptotic p-value
Statistical Analysis 3: Comparison: Developmental Language Disorder; Test type: Other — Accuracy labeling taught verbs in syntactic vs semantic condition (expressive); p = 0.18, Wilcoxon Signed Ranks Test — Asymptotic p-value
Statistical Analysis 4: Comparison: Typical Development; Test type: Other — One-sample Wilcoxon signed rank test with comparison value of 0; p < .001, One-sample Wilcoxon signed rank test — Asymptotic p-value
Statistical Analysis 5: Comparison: Down Syndrome; Test type: Other — One-sample Wilcoxon signed rank test with comparison value of 0; p = 0.034, One-sample Wilcoxon signed rank test — Asymptotic p-value
Statistical Analysis 6: Comparison: Developmental Language Disorder; Test type: Other — One-sample Wilcoxon signed rank test with comparison value of 0; p = 0.063, One-sample Wilcoxon signed rank test — Asymptotic p-value

5. Secondary Outcome: Accuracy Labeling Taught Words - Semantic Condition
Description: After the teaching episodes for the semantic condition participants are asked to label novel verbs expressively. Participants were asked to label each of the 4 taught words per condition one time for a total of 4 trials per condition. This "expressive probe" has a minimum score of 0 and maximum of 4. Higher scores indicate a better outcome.
Time Frame: From date of initial evaluation to focused intervention session, up to 1 month
Population: Analyzed eligible participants
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Typical Development | Down Syndrome | Developmental Language Disorder
Number analyzed (Participants) | 23 | 8 | 7
Score on a scale | 0.52 (0.73) | 1.00 (0.93) | 0.43 (0.79)
Statistical Analysis 1: Comparison: Typical Development; Test type: Other — Accuracy labeling taught verbs in semantic vs combined condition (expressive); p = 0.35, Wilcoxon Signed Ranks Test — Asymptotic p-value
Statistical Analysis 2: Comparison: Down Syndrome; Test type: Other — Accuracy labeling taught verbs in semantic vs combined condition (expressive); p = 0.18, Wilcoxon Signed Ranks Test — Asymptotic p-value
Statistical Analysis 3: Comparison: Developmental Language Disorder; Test type: Other — Accuracy labeling taught verbs in semantic vs combined condition (expressive); p = 0.58, Wilcoxon Signed Ranks Test
Statistical Analysis 4: Comparison: Typical Development; Test type: Other — One-sample Wilcoxon signed rank test with comparison value of 0; p = 0.006, One-sample Wilcoxon signed rank test — Asymptotic p-value
Statistical Analysis 5: Comparison: Down Syndrome; Test type: Other — One-sample Wilcoxon signed rank test with comparison value of 0; p = 0.02, One-sample Wilcoxon signed rank test — Asymptotic p-value
Statistical Analysis 6: Comparison: Developmental Language Disorder; Test type: Other — One-sample Wilcoxon signed rank test with comparison value of 0; p = 0.18, One-sample Wilcoxon signed rank test — Asymptotic p-value

6. Secondary Outcome: Accuracy Labeling Taught Words - Combined Condition
Description: After the teaching episodes for the combined condition participants are asked to label novel verbs expressively. Participants were asked to label each of the 4 taught words per condition one time for a total of 4 trials per condition. This "expressive probe" has a minimum score of 0 and maximum of 4. Higher scores indicate a better outcome
Time Frame: From date of initial evaluation to focused intervention session, up to 1 month
Population: Analyzed eligible participants
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Typical Development | Down Syndrome | Developmental Language Disorder
Number analyzed (Participants) | 23 | 8 | 7
Score on a scale | 0.70 (0.63) | 1.38 (1.41) | 0.71 (1.11)
Statistical Analysis 1: Comparison: Typical Development; Test type: Other — Accuracy labeling taught verbs in syntactic vs combined condition (expressive); p = 0.56, Wilcoxon Signed Ranks Test — Asymptotic p-value
Statistical Analysis 2: Comparison: Down Syndrome; Test type: Other — Accuracy labeling taught verbs in syntactic vs combined condition (expressive); p = 0.10, Wilcoxon Signed Ranks Test — Asymptotic p-value
Statistical Analysis 3: Comparison: Developmental Language Disorder; Test type: Other — Accuracy labeling taught verbs in syntactic vs combined condition (expressive); p = 0.71, Wilcoxon Signed Ranks Test — Asymptotic p-value
Statistical Analysis 4: Comparison: Typical Development; Test type: Other — One-sample Wilcoxon signed rank test with comparison value of 0; p < .001, One-sample Wilcoxon signed rank test — Asymptotic p-value
Statistical Analysis 5: Comparison: Down Syndrome; Test type: Other — One-sample Wilcoxon signed rank test with comparison value of 0; p = 0.024, One-sample Wilcoxon signed rank test — Asymptotic p-value
Statistical Analysis 6: Comparison: Developmental Language Disorder; Test type: Other — One-sample Wilcoxon signed rank test with comparison value of 0; p = 0.10, One-sample Wilcoxon signed rank test — Asymptotic p-value

ADVERSE EVENTS:
Time Frame: Baseline to 30 days
Arm/Group | Typical Development | Down Syndrome | Developmental Language Disorder
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/23 | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT03441685/Prot_SAP_000.pdf